CLINICAL TRIAL: NCT01874522
Title: A Phase 1, Open-label, Randomized, Crossover Study Evaluating the Bioavailability of TAS-102 Tablets Relative to an Oral Solution Containing Equivalent Amounts of FTD and TPI
Brief Title: Study Comparing the Bioavailability of TAS-102 Tablets to an Oral Solution Containing Equivalent Amounts of FTD and TPI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TPU-TAS-102-104
Record Dates: First submitted 2013-06-04; First posted 2013-06-11 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Advanced Solid Tumors (Excluding Breast Cancer)
Keywords: Advanced solid tumors (excluding breast cancer) for which no standard therapy exists
MeSH Terms: interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAS-102 tablets (Experimental)
  Interventions: Drug: TAS-102 tablets
- TAS-102 oral solution (Experimental)
  Interventions: Drug: TAS-102 oral solution

INTERVENTIONS:
Drug: TAS-102 tablets — Crossover bioavailability part: 60 mg/dose, orally, up to 2 single doses separated by 1-week washout.
  Extension part: 35 mg/m2/dose, orally, twice daily on days 1-5 and 8-12 of each 28-day cycle. Number of cycles: until at least one of the discontinuation criteria is met.
  Arms: TAS-102 tablets
Drug: TAS-102 oral solution — 60 mg/dose, orally, up to 2 single doses separated by 1-week washout
  Arms: TAS-102 oral solution

SUMMARY:
The purpose of this study is to compare the bioavailability of TAS-102 tablets to an oral solution containing equivalent amounts FTD and TPI.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, randomized, 2-sequence, 3-period crossover study evaluating the relative bioavailability of TAS-102 tablets compared to an oral solution in patients with advanced solid tumors. This study will be conducted in 2 parts. The crossover bioavailability part will be followed by an extension conducted with TAS-102 tablets only.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent
2. Has advanced solid tumors (excluding breast cancer) for which no standard therapy exists
3. ECOG performance status of 0 or 1
4. Is able to take medications orally
5. Has adequate organ function (bone marrow, kidney and liver)
6. Women of childbearing potential must have a negative pregnancy test and must agree to adequate birth control if conception is possible. Males must agree to adequate birth control.

Exclusion Criteria:

1. Has had certain other recent treatment e.g. anticancer therapy, received investigational agent, within the specified time frames prior to study drug administration
2. Certain serious illnesses or medical condition(s)
3. Has had either partial or total gastrectomy
4. Has unresolved toxicity of greater than or equal to CTCAE Grade 2 attributed to any prior therapies
5. Known sensitivity to TAS-102 or its components
6. Is a pregnant or lactating female
7. Refuses to use an adequate means of contraception (including male patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-07; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Extent of absorption of FTD and TPI following oral administration of TAS 102 tablets or oral solution (Cmax) | Day 1 of Periods 1, 2, and 3
  Pharmacokinetic samples are taken on Day 1 of Periods 1, 2, and 3.
Extent of absorption of FTD and TPI following oral administration of TAS 102 tablets or oral solution (AUC0-last) | Day 1 of Periods 1, 2, and 3
  Pharmacokinetic samples are taken on Day 1 of Periods 1, 2, and 3.
Extent of absorption of FTD and TPI following oral administration of TAS 102 tablets or oral solution (AUC0-inf ) | Day 1 of Periods 1, 2, and 3
  Pharmacokinetic samples are taken on Day 1 of Periods 1, 2, and 3.

SECONDARY OUTCOMES:
Tmax of FTD, TPI, and metabolites of FTD following administration of TAS 102 tablet and oral solution | Day 1 of Periods 1, 2, and 3
  Pharmacokinetic samples are taken on Day 1 of Periods 1, 2, and 3.
T1/2 of FTD, TPI, and metabolites of FTD following administration of TAS 102 tablet and oral solution | Day 1 of Periods 1, 2, and 3
  Pharmacokinetic samples are taken on Day 1 of Periods 1, 2, and 3.
CL/F of FTD and TPI following administration of TAS 102 tablet and oral solution | Day 1 of Periods 1, 2, and 3
  Pharmacokinetic samples are taken on Day 1 of Periods 1, 2, and 3.
Vd/F of FTD and TPI following administration of TAS 102 tablet and oral solution | Day 1 of Periods 1, 2, and 3
  Pharmacokinetic samples are taken on Day 1 of Periods 1, 2, and 3.
Cmax of metabolites of FTD following administration of TAS 102 tablet and oral solution | Day 1 of Periods 1, 2, and 3
  Pharmacokinetic samples are taken on Day 1 of Periods 1, 2, and 3.
AUC0-last of metabolites of FTD following administration of TAS 102 tablet and oral solution | Day 1 of Periods 1, 2, and 3
  Pharmacokinetic samples are taken on Day 1 of Periods 1, 2, and 3.
AUC0-inf of metabolites of FTD following administration of TAS 102 tablet and oral solution | Day 1 of Periods 1, 2, and 3
  Pharmacokinetic samples are taken on Day 1 of Periods 1, 2, and 3.
Safety monitoring including adverse events, vital signs, and laboratory assessments | Through 30 days following last administration of study medication or until initiation of new anticancer treatment
  Standard safety monitoring and grading using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) will be used.
Tumor assessments using Response Evaluation Criteria in Solid Tumors (RECIST) | Every 8 weeks during the extension period through Cycle 6 (ie, through 24 weeks). Thereafter, assessments will be performed at least every 12 weeks according to site standard of care, until at least one of the treatment discontinuation criteria is met.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Von Hoff, MD, Principal Investigator — Scottsdale Healthcare
Locations (1):
- Scottsdale Healthcare, Scottsdale, Arizona, United States